CLINICAL TRIAL: NCT02897271
Title: Demographics, Clinical Characteristics, and Pathology of Eosinophilic Gastritis, Enteritis, and Colitis in a Multi-Site Cohort
Brief Title: Characteristics of Eosinophilic Gastritis, Enteritis, and Colitis in a Multi-Site Cohort
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Office of Rare Diseases (ORD) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2016-4349; 5U54AI117804-03 (NIH)
Record Dates: First submitted 2016-09-02; First posted 2016-09-13 (Estimated); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Eosinophilic Esophagitis; Eosinophilic Gastritis; Eosinophilic Gastroenteritis; Eosinophilic Colitis
Keywords: Eosinophilic Gastrointestinal Disorders
MeSH Terms: conditions — Eosinophilic Esophagitis; Eosinophilic enteropathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to investigate features of patients with Eosinophilic Gastrointestinal Disorders (EGIDs) other than Eosinophilic Esophagitis (EoE) alone, including Eosinophilic Gastritis (EG), Eosinophilic Gastroenteritis (EGE), and Eosinophilic Colitis (EC).

DETAILED DESCRIPTION:
This retrospective chart review study will analyze the demographics, medical history, clinical features, and pathological data of patients with Eosinophilic Gastrointestinal Disorders (EGIDs) other than Eosinophilic Esophagitis (EoE) alone, including Eosinophilic Gastritis (EG), Eosinophilic Gastroenteritis (EGE), and Eosinophilic Colitis (EC).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of an EGID including EG, EGE, and/or EC. Subjects with EoE can be included if they also have another EGID.
* Clinical symptoms of gastrointestinal dysfunction.
* Findings of increased eosinophils on tissue biopsy at the time of diagnosis, before treatment initiated.
* Exclusion of other causes of gastrointestinal eosinophilia.

Exclusion Criteria:

* Gastrointestinal eosinophilia caused by another disorder.
* Diagnosis of EoE without another EGID.
* Insufficient medical record or pathology data available to support an EGID diagnosis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male or female patients of any age with a diagnosis of eosinophilic gastrointestinal disorder (EGID) other than eosinophilic esophagitis (EoE) alone, including eosinophilic gastritis (EG), eosinophilic gastroenteritis (EGE), and eosinophilic colitis (EC).
Sampling Method: Non-Probability Sample
Enrollment: 381 (Actual)
Dates: Start 2016-08; Primary Completion 2019-09 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Mucosal eosinophilia (eos/hpf) | Duration of funding, approximately 5 years
  Mucosal eosinophil levels are measured as eosinophils per high power field (eos/hpf). The primary outcome measure is to determine the change in mucosal eosinophil level (eos/hpf) and to determine if the change in mucosal eosinophil level in eos/hpf correlates with other measures of disease activity.

CONTACTS AND LOCATIONS:
Overall Officials: Marc E Rothenberg, MD, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (6):
- United States (6):
  - University of Arkansas for Medical Science, Little Rock, Arkansas
  - Children's Hospital Colorado, Denver, Colorado
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Rare Diseases Clinical Research Network website — http://www.rarediseasesnetwork.org/cms/CEGIR